CLINICAL TRIAL: NCT04896216
Title: Standardized Patients to Measure and Address Intersectional Stigma: An HIV Prevention Engagement Strategy
Brief Title: Standardized Patients to Measure and Address Intersectional Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006470; R34MH121251 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hiv; HIV Infections; AIDS
Keywords: stigma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stigma Reduction Intervention (Experimental): A Stigma Reduction Intervention curriculum developed using data generated from Stage 1 of the study.
  For stage 2/intervention stage, participants who are providers and randomized to the "Stigma Reduction Intervention" arm through clinic-level randomization
  Interventions: Behavioral: Stigma Reduction Intervention
- Control (No Intervention): For stage 2/intervention stage, participants who are providers and randomized to the "Control" arm through clinic-level randomization

INTERVENTIONS:
Behavioral: Stigma Reduction Intervention — Care providers will complete the Stigma Reduction Intervention curriculum. This study uses a modified Zelen design. Control arm participants will be aware that they are part of an observational study but not that they are in the control arm of an intervention study. This avoids artificially inducing changes to the standards of medical care in facilities randomization to the control arm, a common consequence in RCTs to evaluate population based services.
  Arms: Stigma Reduction Intervention

SUMMARY:
This study aims to develop and evaluate an intervention to reduce enacted stigma in healthcare settings aimed at people living with HIV (PLWH) and men who have sex with men (MSM) in China. Enacted stigma will be measured using a quality of care score collected through unannounced standardized patient (SP) visits to consenting providers in sexual health clinics.

DETAILED DESCRIPTION:
Standardized patients, or trained actors from the community, will conduct a baseline round of unannounced clinic visits with consenting providers for the purposes of observing their clinical performance. SPs will present clinically standardized case scenarios, but the HIV status and sexual orientation of each case will be randomly varied in order to quantify the extent to which HIV stigma and/or homophobia contribute to the deterioration of care quality. Care quality will be calculated using a global score based on a standard checklist administered to SPs following each visit. Results of the baseline visit will inform the development of a stigma reduction intervention for consenting providers employed at clinics randomized to the treatment arm of the study. Design of this intervention has been informed by results of the baseline study and incorporates expert input from members of community advisory boards (CAB), one made up of community members and the other of providers. The intervention will consist of both didactic and skills-building methods and will be delivered both in-person and through follow-up modules online. Didactic portions will include content on topics including clinical management of common STIs, shared decision making, sexual history taking, and working with marginalized populations. Skills-building sessions will include group-based discussion and medical simulation and feedback with trained standardized patients. Follow-up data collection will begin within 2 months of completing the stigma reduction intervention using the same approach as for the baseline data collection. All research activities will take place in Guangzhou, China.

ELIGIBILITY:
Inclusion Criteria:

* Eligible facilities will be those with:

  1. formal government accreditation as a medical center (a basic tenet of all public hospitals in China); and
  2. possession of an accredited on-site laboratory with capacity to provide enzyme-linked immunosorbent assay testing for HIV, treponemal (e.g. Treponema pallidum particle agglutination) and non-treponemal tests (e.g. rapid plasma regain) for syphilis.
* Within eligible and consenting facilities, eligible providers will be those who are licensed at the time of the study to practice dermatovenereology in China.

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kumi Smith, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a baseline study visit, after which treatment arm providers received the training intervention. After the intervention, a follow-up visit was conducted for evaluation purposes. Randomization procedures were conducted at baseline.
Units Other Than Participants: clinics
Groups:
- Stigma Reduction Intervention: Experimental: a stigma reducation training intervention for providers employed at clinics randomized to the intervention arm.
  No intervention: standard of care (i.e. no training intervention)
- Control: Standard of care (i.e. no training intervention)
Period: Overall Study
Arm/Group | Stigma Reduction Intervention | Control
Started | 30; 9 clinics | 29; 8 clinics
Completed | 27; 9 clinics | 18; 7 clinics
Not Completed | 3; 0 clinics | 11; 1 clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stigma Reduction Intervention | Control | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (9) | 43 (9) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 19 | 15 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 25 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MSM Stigma; Domain of Care: Syphilis Testing
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in MSM stigma within each arm (i.e. differences in care quality between men who have sex with men [MSM] vs. straight men). This outcome measures care quality related to whether or not doctors offered a syphilis test.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | 0.078 [-0.079 to 0.235] | 0.034 [-0.181 to 0.248]

2. Primary Outcome: HIV Stigma; Domain of Care: Syphilis Testing
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in HIV stigma within each arm (i.e. differences in care quality between HIV positive vs. HIV negative people). This outcome measures care quality related to whether or not doctors offered a syphilis test.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.201 [-0.406 to 0.005] | 0.034 [-0.181 to 0.248]

3. Primary Outcome: Intersectional Stigma; Domain of Care: Syphilis Testing
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in intersectional stigma within each arm (i.e. differences in care quality between HIV positive MSM vs. HIV negative straight men). This outcome measures care quality related to whether or not doctors offered a syphilis test.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.07 [-0.38 to 0.25] | 0 [0 to 0]

4. Primary Outcome: MSM Stigma; Domain of Care: Diagnostic Effort
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in MSM stigma within each arm (i.e. differences in care quality between men who have sex with men [MSM] vs. straight men). This outcome measures care quality related to the level of diagnostic effort expended by the doctor.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.055 [-0.862 to 0.752] | 0.396 [-0.278 to 1.069]

5. Primary Outcome: HIV Stigma; Domain of Care: Diagnostic Effort
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in HIV stigma within each arm (i.e. differences in care quality between HIV positive vs. HIV negative people). This outcome measures care quality related to the level of diagnostic effort expended by the doctor.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.570 [-1.230 to 0.090] | 0.396 [-0.278 to 1.069]

6. Primary Outcome: Intersectional Stigma; Domain of Care: Diagnostic Effort
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in intersectional stigma within each arm (i.e. differences in care quality between HIV positive MSM vs. HIV negative straight men). This outcome measures care quality related to the level of diagnostic effort expended by the doctor.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | 0.621 [-0.237 to 1.478] | 0.396 [-0.278 to 1.069]

7. Primary Outcome: MSM Stigma; Domain of Care: Patient-centered Care
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in MSM stigma within each arm (i.e. differences in care quality between men who have sex with men [MSM] vs. straight men). This outcome measures care quality related to the patient-centeredness of care provided.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.168 [-0.595 to 0.259] | -0.162 [-0.852 to 0.528]

8. Primary Outcome: HIV Stigma; Domain of Care: Patient-centered Care
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in HIV stigma within each arm (i.e. differences in care quality between HIV positive vs. HIV negative people). This outcome measures care quality related to the patient-centeredness of care provided.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | 0.408 [-0.310 to 1.126] | -0.162 [-0.852 to 0.528]

9. Primary Outcome: Intersectional Stigma; Domain of Care: Patient-centered Care
Description: The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. This outcome quantifies pre-post changes in intersectional stigma within each arm (i.e. differences in care quality between HIV positive MSM vs. HIV negative straight men). This outcome measures care quality related to the patient-centeredness of care provided.
Time Frame: 4 months post-intervention
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Stigma Reduction Intervention | Control
Number analyzed (Participants) | 30 | 25
percentage points | -0.165 [-0.836 to 0.506] | -0.162 [-0.852 to 0.528]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Control: This study uses a modified Zelen design. Control arm participants will be aware that they are part of an observational study but not that they are in the control arm of an intervention study. This avoids artificially inducing changes to the standards of medical care in facilities randomization to the control arm, a common consequence in RCTs to evaluate population based services.
Arm/Group | Stigma Reduction Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT04896216/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04896216/ICF_000.pdf